CLINICAL TRIAL: NCT02129478
Title: Olanzapine for Prevention of Chemotherapy-induced Nausea and Vomiting in Children: A Multi-Centre Feasibility Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Pediatric Oncology Group of Ontario (Other)
Responsible Party: Principal Investigator, Lee Dupuis, Pharmacy Clinical Manager, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1000040306
Record Dates: First submitted 2014-04-28; First posted 2014-05-02 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: olanzapine; pediatrics; chemotherapy-induced nausea; chemotherapy-induced vomiting
MeSH Terms: conditions — Vomiting | interventions — Olanzapine

ARMS (1):
- Olanzapine (Experimental)
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — Patients will receive olanzapine once daily starting just before the first dose of chemotherapy within the study chemotherapy block and continuing until discharge from hospital or for a maximum of 4 doses after the last dose of chemotherapy.
  Olanzapine will be dosed at 0.14mg/kg/dose (maximum 10mg/dose) as a single daily oral dose rounded to the nearest increment of a half-tablet (2.5mg).
  Other Names: Zyprexa

SUMMARY:
Olanzapine is licensed for use in adults in Canada and in teens in the US with mental illness. It is also often used for the management of mental illness in children. This study will describe the feasibility of giving olanzapine plus other usual medications to prevent chemotherapy induced nausea and vomiting (CINV) to 15 children aged 4 to 18 years.

What has been done already? - In adult cancer patients, olanzapine improved the control of CINV. None of the adults studied experienced any serious side effects from olanzapine.

What is being studied and how will the study be conducted? - On each day that chemotherapy is given, olanzapine will be given to 15 children along with their regular medications to prevent CINV. Investigators will study each child only during one chemotherapy cycle. Participants' blood sugar, liver function tests (AST and ALT), prolactin and triglyceride levels, blood pressure, weight, mood and behavior during the time they receive olanzapine will be evaluated to see if they change. Investigators will record anything serious that happens while children receive olanzapine. If any child stops olanzapine early or decides to decrease the dose, the reason will be recorded. Each child and their guardian will record their nausea severity and the times they vomit or retch on each day they receive chemotherapy and for 8 days afterwards.

How will the study help? - This study will help investigators decide if it is feasible to conduct a larger study to find out if olanzapine improves CINV control in children. If most children are able to take olanzapine as set out in the study without having significant side effects, then a larger study would be feasible.

ELIGIBILITY:
Inclusion Criteria:

* 4 to 18 years old
* English-speaking and have an English-speaking parent/guardian
* Have the minimum cognitive ability of a 4 year old as assessed by a health care professional
* Scheduled to receive moderately to highly emetogenic chemotherapy as assessed using the Pediatric Oncology Group of Ontario Guideline for emetogenicity Classification of Antineoplastic Agents in Children on at least one day of a course of chemotherapy
* Scheduled to receive either ondansetron, granisetron or palonosetron with or without dexamethasone on a scheduled basis as ordered by the patient's clinical team as per the usual antiemetic standard of care
* Weigh at least 14kg
* Have serum total bilirubin ≤ 3 mg/dl (50 µmol/L), and ALT and AST ≤ 3x upper limit of normal for age
* Consent to use adequate contraception or remain abstinent on each day olanzapine is given and for 5 days afterward if of child-bearing potential

Exclusion Criteria:

* Brain tumor patients
* Have had treatment within 14 days prior to study enrollment with olanzapine or 30 days prior to study enrollment with another antipsychotic agent
* Planned to receive amifostine, CYP1A2 inducers or inhibitors, other antipsychotic agents or quinolone antibiotics while receiving olanzapine;
* Have uncontrolled hypertension
* Receive other antipsychotic agents, amifostine, citalopram, CYP1A2 inducers or inhibitors, quinolone antibiotics while receiving olanzapine
* Receive scopolamine patches, phenothiazines, acupressure or acupuncture during the study period
* Planned to receive any antiemetic agents other than dexamethasone, ondansetron, granisetron, palonosetron, aprepitant or fosaprepitant on a scheduled basis
* Have a history of neuroleptic malignant syndrome, a seizure disorder, hypersensitivity to olanzapine, cardiac arrhythmias including prolonged QT, low left ventricular ejection fraction, or a history of uncontrolled diabetes mellitus
* Are pregnant or breast-feeding

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2014-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Dupuis, RPh, PhD, Principal Investigator — The Hospital for Sick Children
Locations (3):
- Canada (3):
  - Children's Hospital, London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Result] Flank J, Schechter T, Gibson P, Johnston DL, Orsey AD, Portwine C, Sung L, Dupuis LL. Olanzapine for prevention of chemotherapy-induced nausea and vomiting in children and adolescents: a multi-center, feasibility study. Support Care Cancer. 2018 Feb;26(2):549-555. doi: 10.1007/s00520-017-3864-8. Epub 2017 Aug 30. PMID 28856448
- See also: Link to published study results — http://rdcu.be/vpup

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Olanzapine
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Olanzapine
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 11.1 [4.1 to 17.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 15

OUTCOME MEASURES:

1. Primary Outcome: Patient Outcomes
Description: Our primary study outcome evaluated the feasibility of a future trial of olanzapine that would evaluate the contribution of olanzapine to chemotherapy-induced nausea and vomiting (CINV) control in pediatric oncology patients. A future trial was considered feasible if the following patient outcomes were met: mean time to enroll 15 patients was 12 months or less per site, 12 or more patients took at least half of the planned olanzapine doses, and 3 or less patients experienced significant sedation or dizziness despite dose reduction.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Olanzapine
Number analyzed (Participants) | 15
Participants
  Participants enrolled at 12 months | 15
  Patients taking half olanzapine doses at 12 months | 15
  Patients with sedation or dizziness at half dose | 0

2. Secondary Outcome: Proportion of Patients With Complete CINV Control
Description: The proportion of children achieving complete CINV control (no nausea, vomiting, or retching and no use of breakthrough antiemetic agents) during the acute (24 hours after the last dose of chemotherapy is administered) and delayed phases (the 7 days following the acute phase) will be described. The duration of assessment will depend on the number of days each individual patient receives chemotherapy. Nausea will be assessed using the Pediatric Nausea Assessment Tool (PeNAT).
Time Frame: During the acute (24 hours) and delayed (7 days after acute phase) phases, up to 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Olanzapine
Number analyzed (Participants) | 15
Participants | 0

3. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: All early discontinuation of olanzapine or dose reduction cases will be reported.
Time Frame: Every day for 30 days after the last dose of the study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Olanzapine
Number analyzed (Participants) | 15
Participants
  # patients with reduced dose | 6
  # patients with drug discontinuation | 2

ADVERSE EVENTS:
Arm/Group | Olanzapine
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 8/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine (N=15)
Sedation (Nervous system disorders) | 6 (6)
Blurry vision (Eye disorders) | 1
Increased plasma GGT values (Blood and lymphatic system disorders) | 1
Mild dizziness (General disorders) | 2
Mild orthostatic hypotension (General disorders) | 1
Hypertriglyceridemia (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No